CLINICAL TRIAL: NCT02425020
Title: Effects of Meat Protein Administration on Body Composition, Strength, Muscle Structure and Markers of Muscle Damage and Health in Athletes
Brief Title: Meat and Whey Protein Supplementation in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Responsible Party: Principal Investigator, Fernando Naclerio, Principal Lecturer, University of Greenwich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: uREC0015
Record Dates: First submitted 2015-04-13; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Dietary Modification
Keywords: Supplement; performance; whey; meat; protein
MeSH Terms: interventions — Meat Proteins; Whey Proteins; Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Meat protein (Experimental): Post workout (training days) or breakfast (non training days) 20g of meat protein mixed with 250ml of orange juice and water
  Interventions: Dietary Supplement: Meat Protein
- Whey Protein (Experimental): Post workout (training days) or breakfast (non training days) 20g of whey protein isolate mixed with 250ml of orange juice and water
  Interventions: Dietary Supplement: Whey protein
- Carbohydrate (Active Comparator): Post workout (training days) or breakfast (non training days) maltodextrin mixed with 250ml orange juice and water
  Interventions: Dietary Supplement: Carbohydrate

INTERVENTIONS:
Dietary Supplement: Meat Protein — Immediately (<10 min) after completing each training session (resistance training or sport specific workout), participants will consume a beverage containing 20g of meat protein mixed with 250 ml of orange juice and water. On non-training days supplement will be ingested before breakfast.
  Arms: Meat protein
Dietary Supplement: Whey protein — Immediately (<10 min) after completing each training session (resistance training or sport specific workout), participants will consume a beverage containing 20g of whey protein mixed with 250 ml of orange juice and water. On non-training days supplement will be ingested before breakfast.
  Arms: Whey Protein
Dietary Supplement: Carbohydrate — Immediately (<10 min) after completing each training session (resistance training or sport specific workout), participants will consume a beverage containing about 20g of maltodextrin mixed with 250 ml of orange juice and water. On non-training days supplement will be ingested before breakfast.
  Arms: Carbohydrate

SUMMARY:
The aim of this project is to investigate the potential benefits of combining a new protein meat hydrolysates extract with a regular resistance training programme on (a) body composition (b) performance (c) muscle structure (d) general markers health and immunity in athletes. As a second objective the investigators will analyse potential differences obtained from the ingestion of the new hydrolysates meat protein extract compared to the ingestion of others commercially available protein sources such as whey or casein.

DETAILED DESCRIPTION:
This investigation involves a 8 weeks randomised, balanced, double blind parallel group between-subjects design aimed to analyse the effects of combining exercise and a post exercise nutrition strategy (hydrolysates meat protein, whey protein or a isocaloric only carbohydrate placebo) on training outcomes, markers of immunity and health after a period of regular training and feeding intervention. Participants will be divided in three-treatment groups 1) Hydrolysed meat-protein (MEAT); 2) Whey (W) and 3) non-protein iso-energetic placebo (CHO). Once considered eligible for the study, and after an initial familiarisation period and baseline tests, participants will be randomly assigned to one of the intervention groups: MEAT; W and CHO. Each group will follow a 8-week periodised resistance training intervention combined with one of the three specific supplementation treatments (MEAT, W or CHO). Measurements of general markers of health, immunity, body composition, muscle structure and performance will be determined before and after the training intervention.

Once informed consent and health history have been obtained, after the baseline Assessment (t1), participants will divided into three similar profile groups, matched by body mass, age, sex and performance. 1) The meat protein group (MEAT n=10) that will take 250 ml of orange juice mixed with 20g of hydrolysates meat protein powder and water 2) The whey group (n=10) will take 20 g of whey intact isolate powder mixed with 250 ml of orange juice and water 3) the contrast group (P n=10) that will take an iso-energetic non-protein, only carbohydrate (maltodextrin) placebo.

Participants: Thirty participants, recruited from the University Campus, will take part in the project. After being informed of all risk, discomforts, and benefits involved, participants will sign a written informed consent regarding their participation.

Intervention Familiarization period: Participants will undertake 3 sessions of familiarization (1 weeks). A qualified strength and conditioning coach will control and assists participants in order to guarantee a correct execution of the selected exercise. All participants will be instructed about the appropriate use of the Rate of Perceived Exertion (0-10) scale to control the load and training intensity.

Resistance Training: The resistance-training program will be designed to increase strength and mass of all major muscle groups. The program will be undertaken on three non-consecutive days per week, under the supervision of strength and conditioning coaches, preferable Strength and Conditioning master students. Training workout will be performed during the afternoon (between 3pm and 6pm) with at least 48 hours between sessions.

Each session will begin with individualized warm-up (5-minute warm-up stretches, followed by one set of eight repetitions of six resistance training exercises without any additional weight). Workout will involve 8 resistance exercises per 3 sets of 6 to 10 repetitions at 70% to 85% of an individual 1RM. Exercises will be performed using free-weights, elastic bands, sticks and machines selected to stress the major muscle groups. Resting periods of around 2 min will be allowed sets. Participants will be instructed to maintain the proper execution along the entire training session.

Periodization strategy: The intervention will consist of 8-week periodised resistance training programme that will be divided in 3 blocks: First block (1st to 3th week) using a moderate load intensity of around 70%1RM; Second block (4th to 6th week) where the intensity will increase to >75% to 80% 1RM and the third block (7th to 8th week) where the highest loads (>80 to 85% 1RM) will be used. The Rate of Perceive Exertion (0-10) scale (RPE) will be used to appropriately select the load along the training intervention. Resistance training intervention will be appropriately integrated with the regular sport activity performed by the University athletes along the academic period.

Supplementation protocol: Training days: Immediately (<10 min) after com Non-training days: before breakfast. Supplements and placebo will be provided in powder form and should be mixed with an standardised orange juice and water at the moment of consumption. Supplements and placebo will looks and tastes identical.

Thus, a total of one 20g doses will be administered on daily bases. Participants should ingest a total of 56 doses for a total of 8 weeks of study intervention.

Supplement will be provided in 14 days based by a blind researcher after Participants should return back the empty bag of the supplement/placebo consumed during the previous 14 days period.

ELIGIBILITY:
Inclusion Criteria:

* regularly trained athletes,
* aged 18 to 45 years old,
* minimum 3 months of experience in resistance training exercise,
* volunteers,

Exclusion Criteria:

* any musculoskeletal injuries, metabolic conditions, or diseases;
* use of medications, smoking, and nutritional supplements known to affect physical performance, muscle damage or recovery process (e.g., creatine, whey protein, and amino acids) within 6 weeks prior to the start of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Body composition | 8 weeks
  Fat Free mass and Fat Mass.

SECONDARY OUTCOMES:
Muscle Structure | 8 weeks
  Thickness of biceps brachialis short head and vastus lateralis
Muscle damage marker | 8 weeks
  Creatine Kinase (CK)
Analysis of glycaemia | 8 weeks
Analysis of total cholesterol | 8 weeks
Analysis of HDL, cholesterol | 8 weeks
Analysis of LDL,cholesterol | 8 weeks
Analysis of Aspartate amino transferase | 8 weeks
Analysis of Alanine amino transferase | Pre and post 8 weeks intervention programme
Analysis of Triglycerides | 8 weeks
Analysis of Urea | 8 weeks
Analysis of Uric acid | 8 weeks
Immune system (Analysis of Antimicrobial peptides) | 8 weeks
  Antimicrobial peptides
Maximal Strength performance | 8 weeks
  1RM bench press and 1 RM squat
Power performance (jump test on force plate and maximal power at 50% 1RM bench press) | 8 weeks
  jump test on force plate and maximal power at 50% 1RM bench press

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Naclerio, PhD, Principal Investigator — University of Greenwich